CLINICAL TRIAL: NCT00398892
Title: The Effects of Lipoic Acid on Glycaemic Control in Type 2 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-001543-36
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Glycaemic control; Lipoic acid; Diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- 1 (Other): Crossover - placebo then active
  Interventions: Drug: Lipoic acid
- 2 (Other): Crossover - active then placebo
  Interventions: Drug: Lipoic acid

INTERVENTIONS:
Drug: Lipoic acid — Lipoic acid capsules

SUMMARY:
Hypothesis: that lipoic acid supplements taken orally will improve control of blood sugar levels in people with type 2 diabetes.

This study will recruit 18 people with type 2 diabetes, whose diabetes is currently managed on oral agents. Each subject will then either take placebo for 12 weeks followed by lipoic acid for 12 weeks, or lipoic acid followed by placebo.

A blood test for overall diabetes control will be taken at the start and end of each 12 week period, and the change in control will be compared for lipoic acid vs placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled crossover trial of lipoic acid for glycaemic control in type 2 diabetes.

The trial has 3 phases, each lasting 12 weeks. During phases 1 and 3, subjects take lipoic acid or placebo tablets, the order to be determined by randomization. Phase 2 is a 12-week washout period. The intervention is lipoic acid 200mg daily for 1 week, 400mg daily for the second week, and 600mg daily for weeks 3-12. Equivalent numbers of placebo tablets will be taken during the placebo phase.

The principal outcome measure is change in HbA1c between the start and end of lipoic acid supplementation, by comparison with the same change with placebo.

The secondary outcome measure is change in urine albumin:creatinine ratio over the same periods.

Assessments for safety will include standard adverse events reporting, repeated laboratory measurements throughout the study (blood count, renal and liver function) and hypoglycaemia frequency.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age > 18 years
* Capable of giving informed consent
* Treated with oral antidiabetic agents (not insulin)
* HbA1c 7.0 - 8.5% at last measurement (must be within 6 months of study)
* Most recent HbA1c within 1% of all measurements within preceding year
* Prepared to self-test blood glucose on a regular basis
* Prepared to use contraception during study if of child-bearing potential

Exclusion Criteria:

* Unstable cardiac disease (NYHA class III or IV heart failure, or unstable angina or myocardial infarction within last three months)
* Significant renal or hepatic impairment (creatinine>170 micromol/L, alanine transaminase or alkaline phosphatase > 3x upper limit of normal)
* Other medical condition or treatment likely to affect glycaemic control
* Previous history of significant hypoglycaemia
* Pregnancy
* Involvement in other clinical trial in last three months
* Known or suspected sensitivity to trial products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c change for lipoic acid vs placebo | 12 weeks

SECONDARY OUTCOMES:
Urine ACR change for lipoic acid vs placebo | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James D Walker, Principal Investigator — NHS Lothian - St John's Hospital, Livingston
Locations (1):
- Diabetes Department, St John's Hospital, Livingston, Scotland, United Kingdom